CLINICAL TRIAL: NCT02035709
Title: Phase 4 Study of Postoperative Pain Therapy With Hydromorphone Using Patient-Controlled Target-Controlled Infusion (TCI-PCA) vs. Patient-Controlled Analgesia (PCA) After Elective Cardiac Surgery
Brief Title: Postoperative Pain Therapy With Hydromorphone Using TCI-PCA
Acronym: TCI-PCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCI-PCA-001; 2013-002875-16 (EudraCT Number)
Record Dates: First submitted 2013-12-04; First posted 2014-01-14 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Postoperative Pain
Keywords: Therapy
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCI-PCA (Active Comparator): Intravenous Patient-Controlled Analgesia with Target-Controlled Infusion
  Interventions: Drug: Hydromorphone
- PCA (Active Comparator): Intravenous Patient-Controlled Analgesia
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone is given by PCA or TCI-PCA. The TCI-PCA System steer the hydromorphone infusion pump to achieve plasma concentrations of hydromorphone in predefined increasing steps on patient request and in predefined decreasing steps on lack of patient request within predefined plasma concentration range, lock times and infusion speed.

SUMMARY:
Treatment of postoperative pain with hydromorphone (a strong analgesic) using patient-controlled analgesia with target concentrations in blood compared to conventional patient-controlled analgesia after planed cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 40 and 85 years, both genders
* Scheduled for elective cardiac surgery involving thoracotomy and subsequent ICU stay

Exclusion Criteria:

* Administration of other analgesics or sedatives, if not administered in stable dosage for at least 14 days or if not used for premedication and surgery
* Administration of hydromorphone in the period between screening and surgery
* Severe hepatic or renal impairment in medical history
* BMI ≥35 kg/m²
* ASA ≥4

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Hydromorphone Plasma Concentrations | Day 0 (Visit 2 on day of surgery): -1, 3, 30, 90, 91, 93, 95, 97, 100 min after start of hydromorphone infusion but before extubation; one sample each hour for the following 17 hours after extubation
  Predictive accuracy of the "Erlanger pharmacokinetic model" of hydromorphone administered via TCI, TCI-PCA and conventional PCA during the early postoperative stage

SECONDARY OUTCOMES:
Numerical Rating Score | Day 0 (Visit 2 on day of surgery): -1, 3, 30, 90, 91, 93, 95, 97, 100 min after start of hydromorphone infusion but before extubation; one sample each hour for the following 17 hours after extubation
  Comparison between hydromorphone TCI-PCA and conventional hydromorphone PCA during the early postoperative stage regarding analgetic efficiency

OTHER OUTCOMES:
Amount of Hydromorphone Administered | Day 1 (Visit 3 on first day after surgery)
  Comparison between hydromorphone TCI-PCA and conventional hydromorphone PCA during the early postoperative stage regarding the amount of hydromorphone administered

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jeleazcov, MD, Associate Professor, Principal Investigator — Department of Anesthesiology, University Hospital Erlangen
Locations (2):
- Germany (2):
  - Department of Anesthesiology, University Hospital Erlangen, Erlangen, Bavaria
  - Department of Anesthesiology, University Hospital Erlangen, Erlangen

REFERENCES:
- [Background] Jeleazcov C, Saari TI, Ihmsen H, Mell J, Frohlich K, Krajinovic L, Fechner J, Schuttler J. Population pharmacokinetic modeling of hydromorphone in cardiac surgery patients during postoperative pain therapy. Anesthesiology. 2014 Feb;120(2):378-91. doi: 10.1097/ALN.0b013e3182a76d05. PMID 23958818
- [Derived] Wehrfritz A, Ihmsen H, Fuchte T, Kim M, Kremer S, Weiss A, Schuttler J, Jeleazcov C. Postoperative pain therapy with hydromorphone; comparison of patient-controlled analgesia with target-controlled infusion and standard patient-controlled analgesia: A randomised controlled trial. Eur J Anaesthesiol. 2020 Dec;37(12):1168-1175. doi: 10.1097/EJA.0000000000001360. PMID 33009192
- [Derived] Ihmsen H, Rohde D, Schuttler J, Jeleazcov C. External Validation of a Recently Developed Population Pharmacokinetic Model for Hydromorphone During Postoperative Pain Therapy. Eur J Drug Metab Pharmacokinet. 2017 Feb;42(1):17-28. doi: 10.1007/s13318-015-0318-x. PMID 26797808